CLINICAL TRIAL: NCT01828320
Title: Triple Vulnerability? Circadian Tendency, Sleep Deprivation and Adolescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Allison Harvey, Professor of Clinical Psychology, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01HD071065-01A1 (NIH)
Record Dates: First submitted 2013-04-02; First posted 2013-04-10 (Estimated); Results first posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Eveningness/Sleep
Keywords: Risk: Emotional, Cognitive, Behavioral, Social, Physical
MeSH Terms: conditions — Behavior | interventions — Cognitive Behavioral Therapy; Chronotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment 1 (Experimental): Integrates evidence-based treatments derived from basic research on the circadian system
  Interventions: Behavioral: Cognitive Behavior Therapy for Insomnia, Interpersonal and Social Rhythms Therapy, Chronotherapy
- Treatment 2 (Active Comparator): Psychoeducation on the inter-associations between sleep, diet, exercise and stress.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy for Insomnia, Interpersonal and Social Rhythms Therapy, Chronotherapy
  Arms: Treatment 1
Behavioral: Psychoeducation
  Arms: Treatment 2

SUMMARY:
There is an urgent need to identify modifiable mechanisms contributing to risk and vulnerability among youth. The investigators test the hypothesis that eveningness, the tendency to go to sleep late and wake late, is an important contributor to, and even cause of, vicious cycles that escalate vulnerability and risk among youth. This study seeks to determine whether two interventions to reduce eveningness can reduce risk and confer resilience in critical aspects of health, development and functioning in youth.

DETAILED DESCRIPTION:
Teens who exhibit a circadian tendency toward eveningness ('night-owls') follow a delayed sleep schedule, increasing activity later in the day and both going to sleep and getting up later, compared to morning-types ('larks'). The circadian tendency toward eveningness during adolescence arises from a confluence of psychosocial, behavioral and biological factors and is an important contributor to, and maybe even cause of, vicious cycles that escalate vulnerability and risk for poor health and major forms of psychopathology. Indeed, an evening circadian tendency has been associated with a wide range of adverse effects including poorer health, poorer academic performance, poorer self-regulation, greater use of substances, greater tendency for impulsivity, more depression and anxiety, greater emotional instability and more aggressive and antisocial behavior. While the biological shift toward eveningness during puberty may be difficult to modify, the psychosocial and behavioral contributors are modifiable. Moreover, modifying these contributors will eliminate key factors that exacerbate the biological shift. The proposed research will advance current knowledge on the role of eveningness as a mechanism contributing to poorer outcomes during adolescence. The investigators aim to reduce eveningness among 10-18 year olds via an intervention which integrates evidence-based treatments derived from basic research on the circadian system (Treatment 1) compared to a psychoeducational intervention that highlights the interplay between sleep, diet, exercise and stress (Treatment 2). The investigators will randomly allocate adolescents with an evening circadian tendency, and who are 'at risk' in at least one of five health domains (emotional, cognitive, behavioral, social, physical), to either: (a) Treatment 1 (n = 86) or (b) Treatment 2 (n = 86). Measures will be taken pre-treatment, post-treatment, and at 6 and 12 months post-treatment. This research is a first step within a longer term plan to accelerate knowledge on the potentially powerful positive effects, for the developing neural system, of simple, disseminable psychosocial interventions specifically designed to target modifiable risk factors across adolescence.

ELIGIBILITY:
Inclusion criteria.

1. Scoring within the lowest quartile of the Children's Morningness-Eveningness Preferences Scale (CMEP; 27 or lower) and a 7-day sleep diary showing a sleep onset time of of 10:40 pm or later for 10-13 year olds, 11 pm or later for 14-16 year olds, and 11:20 pm or later for 17-18 year olds at least 3 nights per week. Must have had the current pattern of late bedtimes for the last 3 months.
2. 'At risk' in one of the five health domains: emotional, behavioral, social, physical, and cognitive. Emotional risk will be operationalized as a score of 4 or above on any of the following items on the Child Depression Rating Scale: Difficulty Having Fun, Social Withdrawal, Irritability, Depressed Feelings, Excessive Weeping, or a T-score of 61 or above on the Multidimensional Anxiety Scale for Children (MASC), based on age group (10-11 years, 12-15 year, 16-19 years) using the MASC-10 Profile. Behavioral risk will be operationalized as a Sensation Seeking Scale score greater than 3.93 for males ages 10-13, greater than 3.19 for females 10-13, greater than 4.07 for males 14-18, or greater than 3.19 for females 14-18; taking Attention-deficit/hyperactivity disorder (ADHD) medication or Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children (KSADs) diagnosis of ADHD; current alcohol or substance abuse; or past alcohol or substance dependence. Social and cognitive risk will be defined as "worse" than others the teen's age in one or more social behavior from Child Behavior Checklist (CBCL) Section VI or failing one or more academic class from CBCL Section VII, respectively. Physical risk will be operationalized as a Physical Health Questionnaire-15 score of 4 or above, six or more days of school absences, or a BMI above the 85th percentile for the participant's sex and age.
3. Age between 10 and 18 and living with a parent or guardian and and attending a class/job by 9am at least 3 days per week;
4. English language fluency;
5. Able and willing to give informed assent.

Exclusion criteria.

1. An active, progressive physical illness (e.g., cancer, respiratory disorder) or neurological degenerative disease directly related to the onset and course of the sleep disturbance;
2. Evidence from clinical diagnosis or report by youth or parent of sleep apnea, restless legs or periodic limb movements during sleep. Youth presenting with provisional diagnoses of any of these disorders (e.g., sleep apnea) will be referred for a non-study polysomnography (PSG) evaluation at the parent's discretion and will be enrolled only if the diagnosis is disconfirmed;
3. Mental retardation, autism spectrum disorder, or other significantly impairing pervasive developmental disorder. Based on previous recruitment experiences in our youth depression study, we expect this exclusion to be invoked very infrequently (once every few years);
4. Bipolar disorder or schizophrenia or another current Axis I disorder if there is a significant risk of harm and/or decompensation if treatment of that comorbid condition is delayed as a function of participating in any stage of this study. Otherwise, we will allow all other comorbid psychiatric conditions to (i) to maximize representativeness and (ii) because a byproduct may be that the treatment constitutes a helpful 'transdiagnostic' treatment for youth across psychiatric disorders.
5. A medication-free group may be difficult to recruit and would likely be unrepresentative. Hence, participants will not be excluded on the basis of stable use of medications (> 4 weeks). The exception was use of hypnotics and other medications known to alter sleep (e.g., melatonin).
6. History of substance dependence in the past six months;
7. Current suicide risk sufficient to preclude treatment on an outpatient basis.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 176 (Actual)
Dates: Start 2013-03; Primary Completion 2017-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison G Harvey, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

REFERENCES:
- [Derived] Dong L, Dolsen MR, Martinez AJ, Notsu H, Harvey AG. A transdiagnostic sleep and circadian intervention for adolescents: six-month follow-up of a randomized controlled trial. J Child Psychol Psychiatry. 2020 Jun;61(6):653-661. doi: 10.1111/jcpp.13154. Epub 2019 Nov 26. PMID 31773734
- [Derived] Gumport NB, Dolsen EA, Harvey AG. Usefulness and utilization of treatment elements from the Transdiagnostic Sleep and Circadian Intervention for adolescents with an evening circadian preference. Behav Res Ther. 2019 Dec;123:103504. doi: 10.1016/j.brat.2019.103504. Epub 2019 Nov 1. PMID 31678861
- [Derived] Dong L, Gumport NB, Martinez AJ, Harvey AG. Is improving sleep and circadian problems in adolescence a pathway to improved health? A mediation analysis. J Consult Clin Psychol. 2019 Sep;87(9):757-771. doi: 10.1037/ccp0000423. Epub 2019 Jun 27. PMID 31246052
- [Derived] Harvey AG, Hein K, Dolsen EA, Dong L, Rabe-Hesketh S, Gumport NB, Kanady J, Wyatt JK, Hinshaw SP, Silk JS, Smith RL, Thompson MA, Zannone N, Blum DJ. Modifying the Impact of Eveningness Chronotype ("Night-Owls") in Youth: A Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2018 Oct;57(10):742-754. doi: 10.1016/j.jaac.2018.04.020. Epub 2018 Aug 15. PMID 30274649

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Based in a university clinic, from March 2013 to March 2016, youth were randomly assigned, stratified by sex and age (10-14 years, 15-18 years), in a 1:1 parallel group design, to receive either Transdiagnostic Sleep and Circadian Intervention (TranS-C) or Psychoeducation (PE). Sibling pairs (n = 3) were randomized to the same condition.
Groups:
- Trans-C: Integrates evidence-based treatments derived from basic research on the circadian system
  Cognitive Behavior Therapy for Insomnia, Interpersonal and Social Rhythms Therapy, Chronotherapy
- Psychoeducation: Psychoeducation on the inter-associations between sleep, diet, exercise and stress.
  Psychoeducation
Period: Overall Study
Arm/Group | Trans-C | Psychoeducation
Started | 89 | 87
Received Allocated Intervention | 87 | 86
At Follow-up | 81 | 82
Analyzed | 89 | 87
Completed | 81 | 82
Not Completed | 8 | 5
Not completed — Lost to Follow-up | 1 | 3
Not completed — Withdrawal by Subject | 7 | 2

BASELINE CHARACTERISTICS:
Population: Youth aged 10 to 18 years with an evening chronotype and who were "at risk" in 1 of 5 health domains. Participants included 176 youth recruited through clinicians or advertisements.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trans-C | Psychoeducation | Total
Number analyzed (Participants) | 89 | 87 | 176
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 89 | 87 | 176
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.76 (1.94) | 14.78 (1.74) | 14.77 (1.84)
Sex: Female, Male [Count of Participants; unit: Participants] — Youth aged 10 to 18 years with an evening chronotype and who were"at risk"in 1 of 5 health domains.
  Participants included 176 youth recruited through clinicians or advertisements.
  Participants
    Female | 49 | 53 | 102
    Male | 40 | 34 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 13 | 27
  Not Hispanic or Latino | 75 | 74 | 149
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 11 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 4 | 8 | 12
  White | 58 | 56 | 114
  More than one race | 14 | 16 | 30
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 89 | 87 | 176
Education Level (at baseline) [Count of Participants; unit: Participants]
  Grade 5 | 4 | 1 | 5
  Grade 6 | 4 | 3 | 7
  Grade 7 | 6 | 8 | 14
  Grade 8 | 11 | 14 | 25
  Grade 9 | 16 | 12 | 28
  Grade 10 | 22 | 24 | 46
  Grade 11 | 13 | 12 | 25
  Grade 12 | 12 | 13 | 25
  College | 1 | 0 | 1
Family annual income ($) [Count of Participants; unit: Participants]
  <20,000 | 2 | 4 | 6
  20,001 - 50,000 | 11 | 10 | 21
  50,001 - 100,000 | 26 | 16 | 42
  100,000+ | 47 | 55 | 102
  Refused to answer/missing | 3 | 2 | 5
Any current K-SADS Diagnosis (teen report) [Count of Participants; unit: Participants] — K-SADS = Schedule for Affective Disorders and Schizophrenia for School-Age Children. The K-SADS was administered separately to youth and one parent/caregiver to assess for participant current and lifetime Axis I disorders at the pretreatment assessment. Population: The number analyzed includes only those with data on this variable.
  Participants
    number analyzed (Participants) | 87 | 84 | 171
    (all) | 34 | 29 | 63
Any past K-SADS Diagnosis (teen report) [Count of Participants; unit: Participants] — K-SADS = Schedule for Affective Disorders and Schizophrenia for School-Age Children. The K-SADS was administered separately to youth and one parent/caregiver to assess for participant current and lifetime Axis I disorders at the pretreatment assessment. Population: The number analyzed includes only those with data on this variable.
  Participants
    number analyzed (Participants) | 86 | 85 | 171
    (all) | 40 | 37 | 77
Any current K-SADS Diagnosis (parent report) [Count of Participants; unit: Participants] — K-SADS = Schedule for Affective Disorders and Schizophrenia for School-Age Children. The K-SADS was administered separately to youth and one parent/caregiver to assess for participant current and lifetime Axis I disorders at the pretreatment assessment. Population: The number analyzed includes only those with data on this variable.
  Participants
    number analyzed (Participants) | 85 | 83 | 168
    (all) | 21 | 28 | 49
Any past K-SADS Diagnosis (parent report) [Count of Participants; unit: Participants] — K-SADS = Schedule for Affective Disorders and Schizophrenia for School-Age Children. The K-SADS was administered separately to youth and one parent/caregiver to assess for participant current and lifetime Axis I disorders at the pretreatment assessment. Population: The number analyzed includes only those with data on this variable.
  Participants
    number analyzed (Participants) | 84 | 84 | 168
    (all) | 24 | 31 | 55

OUTCOME MEASURES:

1. Primary Outcome: Total Sleep Time (TST) Average on Weeknights Via Daily Sleep Diary
Description: Total sleep time (TST) average on weeknights via Daily Sleep Diary. Change from baseline to post-treatment. The model provides estimates of the mean pre-post change in the Psychoeducation (PE) condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Minutes | 24.72 [7.81 to 41.63] | 13.02 [-4.03 to 30.07]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.34, Intent-to-treat, multilevel modeling; Using intent-to-treat, multilevel modeling with maximum likelihood estimation with the assumption of missing at random, to examine continuous outcomes; d (effect size) = -0.08

2. Primary Outcome: Average Bedtime on Weeknights Measured Via Daily Sleep Diary
Description: Change in average bedtime on weeknights from pre-treatment to post-treatment measured via Daily Sleep Diary. 24-hour decimal format, where times after midnight are expressed as numbers above 24 (ex. 1:30 am is 25.50). The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
hours | -0.03 [-0.22 to 0.15] | -0.05 [-0.23 to 0.14]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.93, intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; d (effect size) = -0.06

3. Primary Outcome: Morning Eveningness Preference Measured Via Childrens Morningness Eveningness Preference Scale
Description: Morning Eveningness preference measured via Childrens Morningness Eveningness Preference Scale(CMEP). Scores range from 10 (Extreme evening preference) to 43 (Extreme morning preference). The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
score on a scale | 3.89 [2.94 to 4.85] | 2.01 [1.05 to 2.97]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.01, Intent-to-treat, multilevel modeling — Using intent-to-treat, multilevel modeling with maximum likelihood estimation with the assumption of missing at random was used to examine continuous outcomes; d (effect size) = -0.50

4. Primary Outcome: Composite Score for Cognitive Domain
Description: Cognitive composite score reflects cognitive functioning and was calculated by averaging the standardized summary scores from two measures: Attentional Control Scale (ACS) and Youth Social Adjustment Scale-Self Report (YSAS). Summary scores were calculated as 1.)ACS = sum of 20 items rated 1- 4; range: 20-80. Higher scores indicate less attentional control; and 2.) YSAS = sum of 6 school/cognitive-related items rated 1-5; range: 6-30. Higher scores indicate worse school-related impairment.
  Per participant, summary scores from the ACS and YSAS were computed and then standardized.
  The final composite (range -2.12 to 2.39) was calculated as the mean of the two standardized scores. Higher scores indicate greater attentional difficulty and school impairment.
  Change in this composite score from baseline to post treatment is reported below. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
units on a scale | -0.04 [-0.19 to 0.12] | 0.11 [-0.04 to 0.27]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.17, Intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.18

5. Primary Outcome: Composite Score for Behavioral Domain
Description: To assess functioning in the Behavioral domain, a Youth Self-Report Composite Risk Score is calculated by taking the mean of standardized summary scores from two measures: Sensation Seeking Scale for Children (SSS) and the Alcohol and Substance Use-Past 30 days (SU; items include questions on caffeine and energy drinks).
  Summary scores were calculated as 1.) SSS = sum of 8 items, rated 1-5, range: 8-40. Higher scores = greater sensation seeking; and 2.) SU = Sum of 23 items rated 0-7, range 0-161. Higher scores = more frequent use.
  For each participant, summary scores from the SSS and SU subscales were computed and standardized. The final composite (range -1.73 to 3.34) was calculated as the mean of the two standardized scores. Higher composite scores indicate higher impairment Change in this composite score from baseline to post-treatment is reported below. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
units on a scale | 0.02 [-0.07 to 0.11] | 0.08 [-0.01 to 0.17]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.31, Intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.07

6. Primary Outcome: Composite Score for Emotional Domain
Description: Youth Self-Report Composite Score, Emotional functioning domain is calculated by taking the mean of standardized summary scores from two measures: Children's Depression Rating Scale-Revised (CDRS) and the Multidimensional Anxiety Scale for Children (MASC).
  Summary scores were calculated as 1.) CDRS = Sum of 17 items. range 17-113. Higher scores indicate greater depressive symptoms; and 2.) MASC= Sum of 39 items. range 0-117. Higher scores indicate greater anxiety.
  For each participant, summary scores from the CDRS and MASC subscales were first computed and then standardized. The final composite (range -2.10 to 3.60) was calculated as the mean of the two standardized scores from the CDRS and MASC. Higher composite scores indicate greater emotional risk (i.e., more depression and anxiety symptoms).
  Change in this composite score from baseline to post treatment is reported below. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
units on a scale | -0.38 [-0.53 to -0.24] | -0.36 [-0.50 to -0.21]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.80, Intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.001

7. Primary Outcome: Composite Score for Social Domain
Description: Composite Score for Social Domain to assess functioning in the Social domain. Calculated by taking the average of the three subscales (ie, friends, family, romantic relationships) from the Youth Social Adjustment Scale - Self Report.
  Youth Social Adjustment Scale - social items only. 9 items (questions 7-15 out of the 23 item scale), item range 1-5. Summary score is calculated by taking the sum of all 9 items. no reverse coding needed. Summary score range 9-45. Higher score = more impaired adjustment.
  The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: Composite score
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Composite score | -0.04 [-0.17 to 0.09] | -0.03 [-0.17 to 0.10]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.96, Intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.04

8. Primary Outcome: Composite Score for Physical Domain
Description: Composite Score for Physical Domain (physical functioning) is calculated by taking the mean of standardized summary scores from two measures: Modifiable Activity Questionnaire for Adolescents (MAQ) and Physical Health Questionnaire (PHQ).
  Summary scores were calculated as 1.) MAQ = sum of the number of hours per week not active/exercising. Higher scores indicate greater numbers of leisure hours; and 2. PHQ-15 = sum of item (13 items for males, 14 items for females), range 0-30. Higher scores indicate worse somatic complaints.
  For each participant, summary scores from the MAQ and PHQ-15 subscales were first computed and then standardized. The final composite (range -3.95 to 1.86) was calculated as the mean of the two standardized scores. Higher composite scores indicate greater physical health risk.
  Change in this composite score from baseline to post treatment is reported below. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
units on a scale | 0.02 [-0.13 to 0.18] | 0.00 [-0.15 to 0.15]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.83, intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = -0.05

9. Secondary Outcome: Sleepiness Scale
Description: Sleepiness subscale from School Sleep Habits Survey (SSHB). This subscale includes 10 items rated on a 4-point scale (0 - 3), assessing sleepiness. Total scores were calculated by summing all item responses. Possible scores range from 0 to 30, with higher scores indicating greater daytime sleepiness. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment, and to 6-month and 12-month followups
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
units on a scale | -1.33 [-2.28 to -0.37] | 0.26 [-0.67 to 1.19]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.02, Intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.35

10. Secondary Outcome: Dim Light Melatonin Onset
Description: Melatonin levels were measured using 13 saliva samples collected at 30-minute intervals, beginning 5.5 hours before and ending 30 minutes after each participant's average bedtime (computed from 7 nights of sleep diary). For each timepoint (baseline and post-treatment), the dim light melatonin onset (DLMO) was estimated by identifying when melatonin levels crossed the 3.0 pg/ml threshold (i.e., the interpolated time). Change in the interpolated DLMO times from baseline to post treatment (which is an average of 9 weeks after the beginning of treatment) reported. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
hours | -0.01 [-0.02 to 0.00] | 0.01 [0.00 to 0.02]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.04, Intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.28

11. Secondary Outcome: Pittsburgh Sleep Quality Index
Description: Pittsburgh Sleep Quality Index (PSQI). Summary score is calculated by taking the sum of item-level scores. Summary score range 0-21. A higher score means increased severity of difficulty in all sleep area components. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
score on a scale | -1.51 [-2.10 to -0.92] | -0.62 [-1.20 to -0.05]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.04, Intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.29

12. Secondary Outcome: Discrepancy Between Weeknights and Weekends for Total Sleep Time
Description: The discrepancy between weeknights and weekends for Total Sleep Time(TST). The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Minutes | 39.43 [9.03 to 69.84] | -8.67 [-38.74 to 21.40]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.03, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; d (effect size) = -0.44

13. Secondary Outcome: Composite Risk Score of Functioning in Five Health-relevant Domains: Emotional Health (Positivity Ratio)
Description: Composite Risk Score of Functioning in Emotional Health, measured via Ecological Momentary Assessment (EMA), assesses subjective emotional well-being across 7-days, per timepoint using a 9-item short form of the Positive and Negative Affect Scale for Children (PANAS-C), which included 4 positive affect items (min = 4, max = 20; higher scores indicate more positive affect) and 5 negative affect items (min = 5, max = 25; higher scores indicate more negative affect), each rated on a 5-point Likert scale.
  A positivity ratio was calculated by dividing the sum of each affect item scores by the sum of negative affect score per survey day. Higher positivity ratios (range: 0.16-4) indicate higher subjective well-being and less risk.
  Change in average Positivity Ratio from baseline to post treatment (which is an average of 9 weeks after the beginning of treatment) reported. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: ratio
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
ratio | -0.03 [-0.12 to 0.06] | -0.01 [-0.10 to 0.09]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.71, intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.07

14. Secondary Outcome: Child Behavior Checklist: Parent-report Emotional Health Composite Risk Score
Description: Parent Measure. The Emotional Health Composite Risk Score was assessed with a composite score of the Anxious/Depressed and Withdrawn/Depressed subscales of Child Behavior Checklist (CBCL), calculated by taking the mean of standardized summary scores for the items within this domain. This is a parent-reported measure of a teen's emotional health, including items related to anxiety/depression. Range for composite total: 0-42, with higher scores indicating more problems.
  The CBCL Anxious/Depressed subscale is composed of 13-items CBCL items on a scale of 0-2, the range of scores is 0-26, with higher scores indicating more emotional problems.
  The CBCL Withdrawn/Depressed subscale is composed of 8-items CBCL items on a scale of 0-2, the range of scores is 0-16, with higher scores indicating more emotional problems.
  The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition
Time Frame: Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: Composite score
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Composite score | -0.07 [-0.22 to 0.08] | -0.05 [-0.20 to 0.10]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.83, intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.02

15. Secondary Outcome: Discrepancy Between Weeknights and Weekends for Bedtime Via Daily Sleep Diary
Description: The discrepancy between weeknights and weekends for Bedtime(BT) via Daily Sleep Diary. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Minutes | 0.12 [-0.25 to 0.48] | 0.07 [-0.29 to 0.43]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.85, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; d (effect size) = -0.11

16. Secondary Outcome: Discrepancy Between Weeknights and Weekends for Wake Time Via Daily Sleep Diary
Description: The discrepancy between weeknights and weekends for Wake time (WUP) via Daily Sleep Diary. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post-treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Minutes | 0.78 [0.37 to 1.19] | 0.08 [-0.33 to 0.48]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.02, Intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = -0.55

17. Secondary Outcome: Composite Risk Score of Functioning in Five Health-relevant Domains: Cognitive Health
Description: Composite Risk Score of Functioning in Cognitive Health measured via Ecological Momentary Assessment. Participants responded to 11 items that measured their concentration, distractedness, and focus related to their current activity. All items were rated on 5-point Likert scale, where higher scores respectively indicated higher levels of concentration, distractedness, and focus (min = 11, max = 55). The composite risk score was calculated by averaging participant responses over the assessment week. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Measure: Mean (95% Confidence Interval); unit: Composite score
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Composite score | 0.12 [-0.12 to 0.35] | -0.20 [-0.43 to 0.02]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.05, intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = -0.33

18. Secondary Outcome: Composite Risk Score of Functioning in Five Health-relevant Domains: Behavioral Health
Description: Composite Risk Score of Functioning in Behavioral Health measured via Ecological Momentary Assessment was assessed by directly asking participants about eating, drinking, chewing gum, and smoking behavior at the time the phone rang through 6 open-ended EMA questions. Responses were coded. The average weekly frequency of intake of junk food, caffeine, alcohol, nicotine, and other substances was tabulated. The minimum score was 0, and there was no maximum score. Higher scores indicate more risky behaviors and thus more risk. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Measure: Mean (95% Confidence Interval); unit: Composite score
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Composite score | -0.28 [-0.49 to -0.08] | -0.30 [-0.50 to -0.11]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.88, intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.04

19. Secondary Outcome: Composite Risk Score of Functioning in Five Health-relevant Domains: Physical Health
Description: Composite Risk Score of Functioning in Physical Health derived from Ecological Momentary Assessment (EMA). For the physical health domain, responses to a single daily item (e.g., "Were you physically active today?") were used to create a binary score: 1 = active, 2 = inactive. Daily responses were collected over 7 days and both summed (range: 7-14) and averaged for each participant.
  The final composite score reflects the average of these daily values (range: 1 - 2) , where lower scores indicate greater physical activity and lower physical health risk.
  Change in this composite score from baseline to post treatment (which is an average of 9 weeks after the beginning of treatment) is reported below. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
units on a scale | 0.11 [0.04 to 0.19] | 0.11 [0.03 to 0.19]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.97, intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.04

20. Secondary Outcome: Composite Risk Score of Functioning in Five Health-relevant Domains: Social Health
Description: Composite Risk Score of Functioning in Social health measured via Ecological Momentary Assessment was assessed by directly asking participants who the participant was with at the time the phone rang. Participants' responses were then manually coded for companion type on a scale of 0-4. Participants' positivity ratios, as calculated in the Emotional Health (Positivity Ratio) Composite Risk Score of Functioning, were then grouped based on occasions when participants were alone vs. with a family member vs. with a friend vs. other. Positivity ratios within groups were averaged (min = 0.16, max = 4), where higher averages indicated higher subjective well-being and lower risk. The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Measure: Mean (95% Confidence Interval); unit: Composite score
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Composite score
  Social health: Alone | 0.04 [-0.05 to 0.13] | 0.03 [-0.06 to 0.12]
  Social health: With a family member | -0.13 [-0.30 to 0.03] | -0.04 [-0.21 to 0.13]
  Social health: With a peer | 0.12 [-0.16 to 0.41] | 0.06 [-0.31 to 0.20]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Composite Risk Score of Functioning in Social Domain measured via Ecological Momentary Assessment: "Alone"; Test type: Superiority; p = 0.88, intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.01
Statistical Analysis 2: Comparison: Trans-C vs Psychoeducation; Composite Risk Score of Functioning in Social Domain measured via Ecological Momentary Assessment: "With a family member"; Test type: Superiority; p = 0.43, intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = -0.18
Statistical Analysis 3: Comparison: Trans-C vs Psychoeducation; Composite Risk Score of Functioning in Social Domain measured via Ecological Momentary Assessment: "With a peer"; Test type: Superiority; p = 0.37, intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.21

21. Secondary Outcome: Child Behavior Checklist: Parent-report Cognitive Health Composite Risk Score
Description: Parent Measure. Cognitive Health Composite Risk Score was assessed with the Thought Problems and Attention Problems subscale of Child Behavior Checklist (CBCL), calculated by taking the mean of standardized summary scores for the items within this domain. This is a parent-reported measure of a teen's cognitive health, including items related to thought problems. Range for composite total: 0-50, with higher scores indicating more cognitive problems.
  The CBCL Thought Problems subscale is composed of 15-items CBCL items on a scale of 0-2, the range of scores is 0-30, with higher scores indicating more problems.
  The CBCL Attention Problems subscale is composed of 10-items CBCL items on a scale of 0-2, the range of scores is 0-20, with higher scores indicating more problems.
  The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: Composite score
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Composite score | -0.22 [-0.36 to -0.09] | 0.01 [-0.13 to 0.15]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.02, Intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.29

22. Secondary Outcome: Child Behavior Checklist: Parent-report Behavioral Health Composite Risk Score
Description: Parent Measure. The Behavioral Health Composite Risk Score was assessed with a composite score of the Rule-Breaking Behavior and Aggressive Behavior subscales of Child Behavior Checklist (CBCL), calculated by taking the mean of standardized summary scores for the items within this domain. This is a parent-reported measure of a teen's behavioral health, including items related to rule-breaking. Range for composite total: 0-70, with higher scores indicating more behavioral problems.
  The CBCL Rule-Breaking Behavior subscale is composed of 17-items CBCL items on a scale of 0-2, the range of scores is 0-34, with higher scores indicating more rule-breaking behavior.
  The CBCL Aggressive Behavior subscale is composed of 18-items CBCL items on a scale of 0-2, the range of scores is 0-36, with higher scores indicating more aggressive behavior.
  The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: Composite score
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Composite score | -0.07 [-0.22 to 0.08] | 0.01 [-0.15 to 0.16]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.49, intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.07

23. Secondary Outcome: Child Behavior Checklist: Parent-report Social Health Composite Risk Score
Description: Parent Measure. The Social Health Composite Risk Score was assessed with a composite score of the Social Problems subscale of Child Behavior Checklist (CBCL), calculated by taking the mean of standardized summary scores for the items within this domain. This is a parent-reported measure of a teen's social health. The CBCL Social Problems subscale is composed of 11-items CBCL items on a scale of 0-2, the range of scores is 0-22, with higher scores indicating more Social problems.
  The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: Composite score
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Composite score | -0.04 [-0.24 to 0.15] | .03 [-0.16 to 0.22]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.60, intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; d (effect size) = 0.11

24. Secondary Outcome: Child Behavior Checklist: Parent-report Physical Health Composite Risk Score
Description: Parent Measure. The Physical Health Composite Risk Score was assessed with a composite score of the Somatic Complaints subscale of Child Behavior Checklist (CBCL), calculated by taking the mean of standardized summary scores for the items within this domain. This is a parent-reported measure of a teen's Physical health (e.g., "vomiting").
  The CBCL Somatic Complaints subscale is composed of 11-items CBCL items on a scale of 0-2, the range of scores is 0-22, with higher scores indicating more physical problems.
  The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: Composite score
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Composite score | -0.24 [-0.40 to -0.07] | -0.14 [-0.31 to 0.03]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.42, Intent-to-treat, multilevel modeling — [p-value comment as in outcome 3, analysis 1]; d (effect size) = 0.08

25. Secondary Outcome: Child Behavior Checklist: CBCL Sleep Composite
Description: Parent Measure. The Sleep Health Composite Risk Score was assessed with a composite score of sleep from Child Behavior Checklist (CBCL), calculated by taking the mean of standardized summary scores for the items within this domain. This is a parent-reported measure of a teen's sleep health. The CBCL sleep subscale is composed of 7-items CBCL items on a scale of 0-2, the range of scores is 0-14, with higher scores indicating more sleep problems.
  The model provides estimates of the mean pre-post change in the PE condition and the TranS-C condition.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment.
Measure: Mean (95% Confidence Interval); unit: Composite score
Arm/Group | Trans-C | Psychoeducation
Number analyzed (Participants) | 89 | 87
Composite score | -1.43 [-1.83 to -1.03] | -0.67 [-1.07 to -0.26]
Statistical Analysis 1: Comparison: Trans-C vs Psychoeducation; Test type: Superiority; p = 0.01, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; d (effect size) = 0.40

26. Other Pre Specified Outcome: Diagnosis of Psychiatric Disorders
Description: Measured via Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children (KSADS) Interview
Time Frame: Baseline only
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Diagnosis of Sleep Disorders
Description: Measured via Duke Structured Interview for Sleep Disorders
Time Frame: as for outcome 9
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Actigraphy Measured Total Sleep Time
Description: calculated separately for weeknights and weekend nights to also compute the discrepancy between weeknights and weekend nights
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Total Wake Time (TWT)
Description: Actigraphy Measured Sleep Onset Latency (SOL; calculated separately for weeknights and weekend nights) and Wake After Sleep Onset (WASO; calculated separately for weeknights and weekend nights) to create Total Wake Time (SOL+WASO) for weeknights, weekends and to also compute the discrepancy between weeknights and weekend nights
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Actigraphy Measured Daytime Activity Count
Description: calculated separately for weekdays and weekends
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Daily Sleep Diary
Description: total sleep time (weekend nights), weekend night bedtime, weekend rise time, total wake time (SOL+WASO) weeknights, total wake time (SOL+WASO) weekend nights, naps.
Time Frame: as for outcome 9
Reporting Status: Not Posted

32. Other Pre Specified Outcome: "Problems That Are Related to Romantic Relations" Subscale of the Problem Questionnaire
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Internet Behavior Checklist Questionnaire
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Rosenberg Self Esteem Scale Questionnaire
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Rosenberg Self Efficacy Scale Questionnaire
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Sleep Inertia Questionnaire
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Inventory of Parent and Peer Attachment Questionnaire
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

38. Other Pre Specified Outcome: Social Skills Rating Scale Questionnaire
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

39. Other Pre Specified Outcome: Estradiol Hormone Levels
Description: from females only
Time Frame: Baseline only
Reporting Status: Not Posted

40. Other Pre Specified Outcome: Dehydroepiandrosterone (DHEA) Hormone Levels
Description: collected via saliva sample DNA by saliva sample to examine selected circadian and emotion single nucleotide polymorphism (SNP)
Time Frame: Baseline only
Reporting Status: Not Posted

41. Other Pre Specified Outcome: Testosterone Hormone Levels
Description: collected via saliva sample
Time Frame: Baseline only
Reporting Status: Not Posted

42. Other Pre Specified Outcome: Cytokines: Interleukin-6, Tumor Necrosis Factor-α, and C-reactive Protein.
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

43. Other Pre Specified Outcome: Weight (Lbs)
Time Frame: as for outcome 9
Reporting Status: Not Posted

44. Other Pre Specified Outcome: Height (Feet, Inches)
Time Frame: as for outcome 9
Reporting Status: Not Posted

45. Other Pre Specified Outcome: Waist Circumference (cm)
Time Frame: as for outcome 9
Reporting Status: Not Posted

46. Other Pre Specified Outcome: Hip Circumference (cm)
Time Frame: as for outcome 9
Reporting Status: Not Posted

47. Other Pre Specified Outcome: Therapy Process Measure
Description: Credibility Expectancy Questionnaire
Time Frame: Session 2 only
Reporting Status: Not Posted

48. Other Pre Specified Outcome: Emotion "GoNoGo" Task
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

49. Other Pre Specified Outcome: Emotional International Affective Pictures System (IAPS) Task
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

50. Other Pre Specified Outcome: Forward and Backward Digit Span
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

51. Other Pre Specified Outcome: Dimensional Card Sorting Task
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

52. Other Pre Specified Outcome: Food Desire Task and Snack Task (Only a Subsample of Participants)
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

53. Other Pre Specified Outcome: Face Naming Encoding Task (Only a Subsample of Participants)
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

54. Other Pre Specified Outcome: Face Naming Retrieval Task (Only a Subsample of Participants)
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

55. Other Pre Specified Outcome: Flanker Task (Only a Subsample of Participants)
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

56. Other Pre Specified Outcome: Children's Affective Lability Scale
Description: Parent measure
Time Frame: as for outcome 9
Reporting Status: Not Posted

57. Other Pre Specified Outcome: Problems in School Questionnaire
Description: Parent measure
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

58. Other Pre Specified Outcome: Parental Monitoring Questionnaire
Description: Parent measure
Time Frame: Change from baseline to post treatment, which is an average of 9 weeks after the beginning of treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 1 year.
Description: All-cause mortality, Serious, and Other (Not Including Serious) Adverse Events were monitored through occasional assessment and self-report.
Arm/Group | Trans-C | Psychoeducation
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/87
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/87
Other Adverse Events (participants affected / at risk) | 0/89 | 0/87

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT01828320/Prot_SAP_000.pdf